CLINICAL TRIAL: NCT06294509
Title: Feasibility and Effects of Transcutaneous Auricular Vagus Nerve Stimulation Timings in a Sensorimotor Task
Brief Title: TaVNS Application Timing During Robotic Sensorimotor Task
Acronym: SMTaVNS2024
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Olivier Lambercy (Other)
Responsible Party: Sponsor-Investigator, Olivier Lambercy, Adjunct Professor at the Department of Health Sciences and Technology and Co-Director of the Rehabilitation Engineering Laboratory, Swiss Federal Institute of Technology
Organization: Swiss Federal Institute of Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SMTaVNS 2024; 2024-00039 (Registry Identifier: BASEC)
Record Dates: First submitted 2024-02-28; First posted 2024-03-05 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-03

CONDITIONS: Healthy
Keywords: sensorimotor adaptation; motor learning; transcutaneous auricular Vagus nerve stimulation

STUDY DESIGN:
Intervention Model Description: Single-blinded, pseudo-randomised, exploratory, single-centre, national, longitudinal study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- No stimulation (control) (No Intervention): Participants will wear device but will not receive any stimulation
- Movement-unrelated stimulation (control) (Active Comparator): Participants will wear device and receive randomly timed stimulation
  Interventions: Device: in-house developed transcutaneous auricular Vagus Nerve Stimulation device
- pre-movement taVNS (Experimental): Stimulation will start after 500ms of being in the home position, before the onset of the movement cue.
  Interventions: Device: in-house developed transcutaneous auricular Vagus Nerve Stimulation device
- during-movement taVNS (Experimental): Stimulation will occur during the movement phase.
  Interventions: Device: in-house developed transcutaneous auricular Vagus Nerve Stimulation device
- post-movement taVNS (Experimental): Stimulation will occur immediately after a successful trial (no stimulation if the trial is failed).
  Interventions: Device: in-house developed transcutaneous auricular Vagus Nerve Stimulation device

INTERVENTIONS:
Device: in-house developed transcutaneous auricular Vagus Nerve Stimulation device — taVNS in this study involves short electric pulses (0.25 ms) delivered to the ear's skin to activate the auricular branch of the Vagus. The pulses are current-controlled to ensure stability and delivered in a bipolar fashion to prevent skin irritation. Before each session, taVNS is calibrated for each participant. Starting at 0.1 mA, the intensity is increased stepwise until a comfortable maximum (typically 1.5-2.5 mA) is reached. Stimuli are delivered in short trains lasting 0.5 seconds each, with 13 pulses (0.25ms each) per train. Participants receive a maximum of 150 stimuli per session, totaling a maximum of 75 seconds of cumulative stimulation. Participants adapt their movements over up to six sessions across two weeks. The robotic task facilitates accurate movement tracking and provides interactive real-time feedback.
  Arms: Movement-unrelated stimulation (control); during-movement taVNS; post-movement taVNS; pre-movement taVNS

SUMMARY:
The goal of this clinical trial is to evaluate the feasibility and effectiveness of transcutaneous auricular vagus nerve stimulation (taVNS) in enhancing sensorimotor learning and adaptation. This study will focus on healthy individuals performing a robotic sensorimotor task.

Main Questions it Aims to Answer:

How does taVNS, with different timing protocols, affect the feasibility and effectiveness of performing a robotic sensorimotor task? What is the impact of taVNS on sensorimotor learning and adaptation?

Participants Will:

Be pseudo-randomly assigned to one of five experimental groups with different taVNS stimulation timings.

Perform a sensorimotor task multiple times across sessions, spanning a maximum of two weeks or until achieving 70% accuracy in two successive sessions.

Have kinematic data collected by a robot during the task. Have physiological data measured using external sensors. Fill out questionnaires about the feasibility of taVNS and other subjective measures after each session.

Comparison Group:

Researchers will compare the four experimental groups to each other to see if different taVNS stimulation timings affect sensorimotor learning outcomes, as well as to a control group that will receive no stimulation.

DETAILED DESCRIPTION:
Overview:

This study focuses on the potential of transcutaneous auricular Vagus Nerve Stimulation (taVNS) in motor neurorehabilitation for conditions like Parkinson's disease, traumatic brain injury, spinal cord injury, and stroke. taVNS, approved for various neurological conditions and known for its safety, activates neuromodulators contributing to plasticity and motor learning. However, the optimal stimulation parameters, especially timing during movement, are not fully explored.

Study Goals:

Primary Objective: To assess the feasibility and effects of different taVNS timing protocols in a robotic sensorimotor task on sensorimotor learning and adaptation. The hypothesis is that varying taVNS-movement timings will influence both subjective and objective feasibility measures and sensorimotor adaptation.

Secondary Objectives: To compare movement kinematics and contrast perceived stimulation effects with measured physiological outcomes and task performance metrics.

Methodology:

The study will be conducted at Swiss Federal Institute of Technology (ETH) Zurich with healthy subjects using a robotic sensorimotor task to evaluate the feasibility of movement-timed taVNS and its influence on learning new sensorimotor skills.

Participants will be assigned different stimulation timings, with the study assessing motor learning and performance consistency across a maximum of 6 sessions or until 70% success is reached in two successive sessions.

The study design is single-blinded, pseudo-randomized, exploratory, and longitudinal, employing controls like no stimulation and randomly-timed stimulation.

Intervention Details:

Before each session, two electrodes (e.g. TensCare pads) will be connected to the pulse generator and 1) placed on the cymbae conchae of the ear and 2) on the tragus of the ear, allowing for a previously described taVNS biphasic pulse train to travel. Here, biphasic square pulses of 250ms width are sent at 25 Hertz (Hz) frequency for 0.5s at a maximum aptitude of 3 milliamperes (mA). The stimulation pulses are current-controlled, limited to 50 Volts (V) and regulated by a pulse generator that limits deliverable current in hardware by design with serial resistors and diodes.

At the start of the session, participants will use a python graphical user interface (GUI) to calibrate the desired taVNS amplitude by gradually increasing it from minimal 0.1 mA up to the maximal tolerated amplitude below 3 mA in the intervals of 0.1 mA. The level of intensity will be set to 90% of the maximally tolerated amplitude for the person (typical ~1.5-2 mA & limited to 3mA, which is significantly below the safety limit of 50mA (according to the Product Safety Standards for Medical Devices, IEC 60601-2-10:2012). This procedure takes 1-2 min. Following the calibration, the session with the sensorimotor task will begin.

Sensorimotor task The sensorimotor task utilizes a commercial haptic end effector (Touch, 3D systems), a custom made 3D printed handle and a virtual reality environment, implemented in python and PsychoPy software on a Microsoft Windows laptop. The robotic manipulandum is synchronized to a 1cm circular cursor in the workspace of the virtual environment. Additionally, an arm-support (SaeboMas Mini) is used to support the arm against gravity to reduce fatigue and keep the arm in the correct position - elbow is 90 degrees perpendicular to the ground.

The goal of the sensorimotor task is to reach a 2.4cm target at a distance of 10 cm away from a starting position, both visually represented in the virtual environment. In order to successfully complete a trial the participant must reach the target within a time constraint of 0.5 s +/- 0.067 s. There will be a 0.5 s tone sound notifying the target duration of the movement. During this movement the cursor position is hidden and not displayed on the screen (in perturbation and retention phases) in order to force feedforward motor adaptation, rather than visually-guided feedback control, as feedforward adaptation may be impaired in stroke patients. Results of each trial are displayed as 3 distinct possibilities - correct, target reached too quickly, or target not reached. The subject will be notified of the outcome of the trial by the target turning either, green, orange or red respectively. Afterwards the start location will be displayed for the participant to return to. After 1-3 s within the starting point a new trial will be initiated.

Participants will perform 75 baseline trials (no visuomotor rotation) to get familiar with the robotic manipulandum and the environment. Then participants will perform an additional 150 trials in the challenged condition with a virtual rotational field (visuomotor rotation/perturbation), displayed on the screen. Subjects will not be informed about the nature of the sensorimotor challenge and will have to progressively learn the corrective mapping to adapt to the perturbation. No external forces will be applied and the haptic end-effector is solely used to measure handle end-point kinematics. Then subjects will perform 50 trials of the same baseline trials (wash-out) and finally 50 more trials of the rotational field (retention). The time requirement is expected to be 5-10 min for the setup and explanations and ~30 min for the sensorimotor task. Data from each trial will be stored containing the position of the cursor, success/fail and time information for subsequent analysis. Additional movement kinematic data may be collected using inertial measurement unit (IMU) sensors worn on the wrist. The IMU records acceleration and gyroscope measurements and logs data to the experimental computer at a rate of 120Hz. Additionally all data pertaining to stimulation will be stored, this includes timing, impedance measurements and all communication commands to and from the stimulator.

Research Significance:

The findings could inform future clinical studies in neurorehabilitation. The study uses a "Touch™" haptic device for the task, ensuring participant safety and comfort.

Potential side effects of taVNS are minimal and closely monitored.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants above 18 years of age and able to provide informed consent and understand the study requirements

Exclusion Criteria:

* Individuals with major untreated depression, major cognitive and/or communication deficits, and major comprehension and/or memory deficits that may interfere with the informed consent process, task-specific practice, or communication of adverse events will be excluded from the study.
* Neurological conditions such as epilepsy, participation in any other research trial, pregnancy, use of implanted electrical devices, and use of medication or procedure that interferes with vagal functions.
* Pregnancy or trying to get pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Subjectively perceived tolerance of taVNS and perceived difficulty of motor task | From enrollment to end of study at 2 weeks
  The subjective perceived feasibility of the taVNS stimulation paradigm, perceived difficulty level of the task, assessed by an unvalidated questionnaire on the Likert scale.
Success of the sensorimotor challenge | After the intervention
  Measured as % of trials where the end-point reaching target (2.4 cm diameter) was reached within an allocated time period (0.5 s +/- 0.067 s).
Mean Change from Baseline in Galvanic Skin Response (GSR) | During and immediately after taVNS
  Physiological dose response to the taVNS using GSR as indicator
Mean Change from Baseline in Heart Rate (HR) | During and immediately after taVNS
  Physiological dose response to the taVNS using HR as indicator
Mean Change from Baseline in Pupil Diameter (PD) | During and immediately after taVNS
  Physiological dose response to the taVNS using PD as indicator
Mean Change from Baseline in electroencephalogram (EEG) | During and immediately after taVNS
  Physiological dose response to the taVNS using EEG as indicator

SECONDARY OUTCOMES:
Subjectively perceived positive effects of taVNS on motor performance | After each session, from enrollment to end of treatment at 2 weeks
  Subjectively perceived success during taVNS and perceived effects of the taVNS stimulation during the task, assessed by an unvalidated questionnaire on the Likert scale.
Change of movement parameters from baseline | After each session, from enrollment to end of study at 2 weeks
  Movement kinematics, as recorded by robotic sensors, will be analyzed to assess quantitative properties of the movements. For example, mean velocity, smoothness of acceleration and trajectory
Associations between outcomes | upon completion of study, at 2 weeks
  Association between subjective and objective feasibility measures will be analyzed using multiple way ANOVA tests for each of the measures

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
Not planned

REFERENCES:
- [Background] Kim AY, Marduy A, de Melo PS, Gianlorenco AC, Kim CK, Choi H, Song JJ, Fregni F. Safety of transcutaneous auricular vagus nerve stimulation (taVNS): a systematic review and meta-analysis. Sci Rep. 2022 Dec 21;12(1):22055. doi: 10.1038/s41598-022-25864-1. PMID 36543841
- [Background] Baig SS, Kamarova M, Bell SM, Ali AN, Su L, Dimairo M, Dawson J, Redgrave JN, Majid A. tVNS in Stroke: A Narrative Review on the Current State and the Future. Stroke. 2023 Oct;54(10):2676-2687. doi: 10.1161/STROKEAHA.123.043414. Epub 2023 Aug 30. PMID 37646161
- [Background] Badran BW, Peng X, Baker-Vogel B, Hutchison S, Finetto P, Rishe K, Fortune A, Kitchens E, O'Leary GH, Short A, Finetto C, Woodbury ML, Kautz S. Motor Activated Auricular Vagus Nerve Stimulation as a Potential Neuromodulation Approach for Post-Stroke Motor Rehabilitation: A Pilot Study. Neurorehabil Neural Repair. 2023 Jun;37(6):374-383. doi: 10.1177/15459683231173357. Epub 2023 May 20. PMID 37209010
- [Background] Branscheidt M, Hadjiosif AM, Anaya MA, Keller J, Widmer M, Runnalls KD, Luft AR, Bastian AJ, Krakauer JW, Celnik PA. Reinforcement Learning Is Impaired in the Sub-acute Post-stroke Period. bioRxiv [Preprint]. 2023 Jan 25:2023.01.25.525408. doi: 10.1101/2023.01.25.525408. PMID 36747674
- [Background] Dietrich S, Smith J, Scherzinger C, Hofmann-Preiss K, Freitag T, Eisenkolb A, Ringler R. A novel transcutaneous vagus nerve stimulation leads to brainstem and cerebral activations measured by functional MRI. Biomed Tech (Berl). 2008 Jun;53(3):104-11. doi: 10.1515/BMT.2008.022. PMID 18601618
- [Background] Breton-Provencher V, Drummond GT, Sur M. Locus Coeruleus Norepinephrine in Learned Behavior: Anatomical Modularity and Spatiotemporal Integration in Targets. Front Neural Circuits. 2021 Jun 7;15:638007. doi: 10.3389/fncir.2021.638007. eCollection 2021. PMID 34163331
- [Background] Gielow MR, Zaborszky L. The Input-Output Relationship of the Cholinergic Basal Forebrain. Cell Rep. 2017 Feb 14;18(7):1817-1830. doi: 10.1016/j.celrep.2017.01.060. PMID 28199851
- [Background] Izawa J, Shadmehr R. Learning from sensory and reward prediction errors during motor adaptation. PLoS Comput Biol. 2011 Mar;7(3):e1002012. doi: 10.1371/journal.pcbi.1002012. Epub 2011 Mar 10. PMID 21423711
- [Background] Morrison RA, Hulsey DR, Adcock KS, Rennaker RL 2nd, Kilgard MP, Hays SA. Vagus nerve stimulation intensity influences motor cortex plasticity. Brain Stimul. 2019 Mar-Apr;12(2):256-262. doi: 10.1016/j.brs.2018.10.017. Epub 2018 Nov 3. PMID 30409712
- [Background] Rodenkirch C, Carmel JB, Wang Q. Rapid Effects of Vagus Nerve Stimulation on Sensory Processing Through Activation of Neuromodulatory Systems. Front Neurosci. 2022 Jul 5;16:922424. doi: 10.3389/fnins.2022.922424. eCollection 2022. PMID 35864985
- [Background] Bowles S, Hickman J, Peng X, Williamson WR, Huang R, Washington K, Donegan D, Welle CG. Vagus nerve stimulation drives selective circuit modulation through cholinergic reinforcement. Neuron. 2022 Sep 7;110(17):2867-2885.e7. doi: 10.1016/j.neuron.2022.06.017. Epub 2022 Jul 19. PMID 35858623
- [Background] Donegan D, Kanzler CM, Buscher J, Viskaitis P, Bracey EF, Lambercy O, Burdakov D. Hypothalamic Control of Forelimb Motor Adaptation. J Neurosci. 2022 Aug 10;42(32):6243-6257. doi: 10.1523/JNEUROSCI.0705-22.2022. Epub 2022 Jul 5. PMID 35790405
- [Background] Wickens JR, Reynolds JN, Hyland BI. Neural mechanisms of reward-related motor learning. Curr Opin Neurobiol. 2003 Dec;13(6):685-90. doi: 10.1016/j.conb.2003.10.013. PMID 14662369
- [Background] Donegan D, Peleg-Raibstein D, Lambercy O, Burdakov D. Anticipatory countering of motor challenges by premovement activation of orexin neurons. PNAS Nexus. 2022 Oct 25;1(5):pgac240. doi: 10.1093/pnasnexus/pgac240. eCollection 2022 Nov. PMID 36712356
- [Background] Kanzler CM, Averta G, Schwarz A, Held JPO, Gassert R, Bicchi A, Santello M, Lambercy O, Bianchi M. A low-dimensional representation of arm movements and hand grip forces in post-stroke individuals. Sci Rep. 2022 May 9;12(1):7601. doi: 10.1038/s41598-022-11806-4. PMID 35534629
- [Background] Lerman I, Davis B, Huang M, Huang C, Sorkin L, Proudfoot J, Zhong E, Kimball D, Rao R, Simon B, Spadoni A, Strigo I, Baker DG, Simmons AN. Noninvasive vagus nerve stimulation alters neural response and physiological autonomic tone to noxious thermal challenge. PLoS One. 2019 Feb 13;14(2):e0201212. doi: 10.1371/journal.pone.0201212. eCollection 2019. PMID 30759089
- [Background] Mridha Z, de Gee JW, Shi Y, Alkashgari R, Williams J, Suminski A, Ward MP, Zhang W, McGinley MJ. Graded recruitment of pupil-linked neuromodulation by parametric stimulation of the vagus nerve. Nat Commun. 2021 Mar 9;12(1):1539. doi: 10.1038/s41467-021-21730-2. PMID 33750784
- [Background] Machetanz K, Berelidze L, Guggenberger R, Gharabaghi A. Transcutaneous auricular vagus nerve stimulation and heart rate variability: Analysis of parameters and targets. Auton Neurosci. 2021 Dec;236:102894. doi: 10.1016/j.autneu.2021.102894. Epub 2021 Oct 12. PMID 34662844
- [Background] Lloyd B, Wurm F, de Kleijn R, Nieuwenhuis S. Short-term transcutaneous vagus nerve stimulation increases pupil size but does not affect EEG alpha power: A replication of Sharon et al. (2021, Journal of Neuroscience). Brain Stimul. 2023 Jul-Aug;16(4):1001-1008. doi: 10.1016/j.brs.2023.06.010. Epub 2023 Jun 20. PMID 37348704
- [Background] Rong P, Liu J, Wang L, Liu R, Fang J, Zhao J, Zhao Y, Wang H, Vangel M, Sun S, Ben H, Park J, Li S, Meng H, Zhu B, Kong J. Effect of transcutaneous auricular vagus nerve stimulation on major depressive disorder: A nonrandomized controlled pilot study. J Affect Disord. 2016 May;195:172-9. doi: 10.1016/j.jad.2016.02.031. Epub 2016 Feb 10. PMID 26896810
- [Background] Badran BW, Yu AB, Adair D, Mappin G, DeVries WH, Jenkins DD, George MS, Bikson M. Laboratory Administration of Transcutaneous Auricular Vagus Nerve Stimulation (taVNS): Technique, Targeting, and Considerations. J Vis Exp. 2019 Jan 7;(143):10.3791/58984. doi: 10.3791/58984. PMID 30663712
- [Background] Kaniusas E, Kampusch S, Tittgemeyer M, Panetsos F, Gines RF, Papa M, Kiss A, Podesser B, Cassara AM, Tanghe E, Samoudi AM, Tarnaud T, Joseph W, Marozas V, Lukosevicius A, Istuk N, Lechner S, Klonowski W, Varoneckas G, Szeles JC, Sarolic A. Current Directions in the Auricular Vagus Nerve Stimulation II - An Engineering Perspective. Front Neurosci. 2019 Jul 24;13:772. doi: 10.3389/fnins.2019.00772. eCollection 2019. PMID 31396044
- [Background] Dabiri B, Zeiner K, Nativel A, Kaniusas E. Auricular vagus nerve stimulator for closed-loop biofeedback-based operation. Analog Integr Circuits Signal Process. 2022;112(2):237-246. doi: 10.1007/s10470-022-02037-8. Epub 2022 May 10. PMID 35571976
- [Background] Joshi S, Li Y, Kalwani RM, Gold JI. Relationships between Pupil Diameter and Neuronal Activity in the Locus Coeruleus, Colliculi, and Cingulate Cortex. Neuron. 2016 Jan 6;89(1):221-34. doi: 10.1016/j.neuron.2015.11.028. Epub 2015 Dec 17. PMID 26711118